CLINICAL TRIAL: NCT06129812
Title: An Exploration of Candidates for Neoadjuvant Treatment in Resectable Pancreatic Cancer According to Tumor-vessel Relationship and CA 19-9 Levels
Brief Title: An Exploration of Candidates for Neoadjuvant Treatment in Resectable Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NAT in resectable PDAC
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer; Neoadjuvant
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- resectable PDAC with no contact to major vessels (R-no contact)
  Interventions: Drug: Neoadjuvant treatment
- resectable PDAC with contact PV/SMV of ≤180° (R-contact)
  Interventions: Drug: Neoadjuvant treatment
- borderline resectable PDAC with PV/SMV contact >180° and without arterial involvement (BR-V)
  Interventions: Drug: Neoadjuvant treatment

INTERVENTIONS:
Drug: Neoadjuvant treatment — Intravenous gemcitabine-based combination regimens or FOLFIRINOX were included in NAC.

SUMMARY:
An Exploration of Candidates for Neoadjuvant Treatment in Resectable Pancreatic Cancer

DETAILED DESCRIPTION:
The 1,132 patients with resectable or borderline resectable PDAC who underwent surgery between 2007 and 2021 were retrospectively reviewed. Patients with resectable PDAC without contact of major vessels (R-no contact) (n=651), with contact of portal vein or superior mesenteric vein (PV/SMV) ≤180° (R-contact) (n=306), and borderline resectable PDAC without arterial involvement (BR-V) (n=175) were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with resectable or borderline resectable pancreatic ductal adenocarcinoma (PDAC)
* Between January 2007 and June 2021 at Seoul National University Hospital

Exclusion Criteria:

* Patients who had borderline resectable PDAC with arterial invasion
* Patients who received chemotherapy as initial treatment and did not undergo surgery
* Incomplete follow-up data for analysis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients with resectable or borderline resectable pancreatic ductal adenocarcinoma (PDAC)
Sampling Method: Non-Probability Sample
Enrollment: 1132 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date when biopsy results came out until the date of death from any cause or the date of the last visit, whichever came first, assessed up to 60 months
  the time from diagnosis to death from any cause or the date of the last visit

IPD SHARING:
Plan to Share IPD: No